CLINICAL TRIAL: NCT04365335
Title: Stress Biomarkers Leading to Professional Burnout Among People Involved in a Mobile Intensive Care Unit During the COVID-19 Pandemic
Acronym: AUTONOMIC
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-COVID19-11; 2020-A01058-31 (Other: IDRCB)
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Occupational Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assessment of work-related stress — Assessment of burnout, mindfulness, interoceptive awareness, anxiety, post-traumatic stress disorder, coping flexibility and sleep through questionnaires.
Biological: Saliva sample collection — Saliva sample is collected before and after emotional stimulation in order to measure resting-state allostatic load biomarkers: DHEA, cortisol and chromogranine A levels
Other: Cardiac and electrodermal recordings — Electrocardiogram and electrodermal activity (tonic and phasic) is collected at rest and after emotional stimulation.
Behavioral: Assessment of behavioral response to emotional stimulation — Emotional stimulation involves asking the participants to remember a recent event related to the COVID-19 crisis that has been emotionally difficult for them.
  Perceived stress, situational awareness and emotions is assessed after emotional stimulation through questionnaires.

SUMMARY:
This study is aiming at investigating whether professional burnout in people involved in the mobile intensive care unit (in French: Element Mobile de Réanimation, EMR) in Mulhouse (France) can be predicted upstream by a low mindfulness level (as a protective factor) or by a dysregulation of stress pathways with a high level of perceived stress towards an emotional event (psychological index of allostatic load), i.e. an early and silent dysfunctional physiological response (measured by the electrophysiological and biological measurements of allostasis load and parasympathetic brake).

It is part of a global approach aiming at identifying levers to prevent the allostatic load of occupational stress related to large-scale health crises.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer staff member of the Mulhouse mobile intensive care unit (in French: Elément mobile de réanimation, EMR), including military reservists.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to a legal protection measure or unable of giving consent
* Intercurrent pathology with inability to work
* History of psychiatric disorder or cardiac pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of people who have been deployed to serve at the mobile intensive care unit in Mulhouse (France) during the Covid-19 crisis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Professional burnout | 21 days after enrollment (Day 21)
  Professional burnout is measured at D21 by the Burnout Measure Short Version (BMS) questionnaire It is a 10-item questionnaire used to assess burnout regardless of the occupational category.
  Each item is rated from 0 to 6 ("never" to "always"). An average score (sum/10) below 2.4 indicates a very low degree of burnout exposure; a score between 2.5 and 3.4 indicates a low degree of burnout exposure; a score between 3.5 and 4.4 indicates the presence of burnout; a score between 4.5 and 5.4 indicates a high degree of burnout exposure; a score above 5.5 indicates a very high degree of burnout exposure.
Mindfulness level | Day 1
  Mindfulness level is assessed at D0 thanks to the Freiburg Mindfulness Inventory.
  It is a 14 item scale. Each item is rated from 1 to 4 ("almost never" to "almost always"). The total score is between 14 and 56. The mean value in a population of young adults under 36 years of age is 38.5 (+/- 5.1 standard deviation).

SECONDARY OUTCOMES:
Perceived stress level following the emotional stimulation | Day 1
  Perceived stress level is assessed with the Perceived Stress Scale (PSS). It is a 14 item scale. Each item is rated from 0 to 5 ("never" to "very often"). The total score ranges from 0 to 56 with higher scores indicating greater perceived stress.
Parasympathetic flexibility evolution during emotional recall | Day 1
  Parasympathetic flexibility is assessed through dynamic electro-physiological analysis of cardiac and electrodermal conductance recordings.
  Physiological and cognitive reserve of emotional regulation is assessed through the analysis of the spectral power of the 0.1 Hz frequency band at emotional recall.
Sympathetic tone at rest | Day 1
  The activity of the sympathetic tone is assessed by the measurement of the resting state salivary Chromogranin A.
  Physiological and cognitive reserve of emotional regulation is assessed through the analysis of the spectral power of the 0.1 Hz frequency band at emotional recall.
  The activity of the sympathetic tone is assessed by the measurement of the resting salivary Chromogranin A.
Corticotropic activation at rest | Day 1
  Corticotropic activation at rest is assessed through the DHEA/cortisol level ratio
Mood disorders (anxiety / depression) | Day 1
  The Hospital Anxiety and Depression Scale (HAD-s32) is used to assess mood disorders in the general non-psychiatric population. It is used to discriminate between anxiety and depression. Scores greater than 11 are indicative of charcaterized anxiety/depression.
Post-traumatic stress disorder | Day 1
  Post-traumatic disorder is assessed with the PCL-5. It is a 20-item self-administered questionnaire representing DSM-5 PTSD diagnosis symptoms rated by the subject on a scale from 0 ("not at all") to 4 ("extremely") during the past month. Scores range from 0 to 80. A score greater than of 33 evokes the presence of post-traumatic stress disorder.
Sleep quality | Day 1
  Sleep quality is assesses thanks to the Leeds Sleep Evaluation questionnaire (LEEDS). It consists of ten visual analogue scales assessing four aspects of sleep: (i) quality of falling asleep and degree of drowsiness, (ii) quality of sleep, (iii) quality of wakefulness, and (iv) quality of post-wakefulness and performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Elément Militaire de Réanimation (EMR), Mulhouse, France